CLINICAL TRIAL: NCT02305953
Title: Correlation Between Serum Levels of Cytokines and a Chemokine and Vascular Inflammation in Patients With Moderate to Severe Psoriasis
Brief Title: Cytokines and Vascular Inflammation in Psoriasis
Status: Completed | Type: Observational
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: Inno-6037
Record Dates: First submitted 2014-10-31; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Vascular Inflammation; Psoriasis; Coronary Atherosclerosis
Keywords: Psoriasis; Vascular Inflammation; Coronary Atherosclerosis; Ascending aorta; PET scan; Cytokine; Chemokine
MeSH Terms: conditions — Psoriasis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Frozen serum: The cohort consists of original subjects from the Inno-6025 Trial who previously consented to measuring protein in the blood involved in skin inflammation.

SUMMARY:
Psoriasis is an inflammatory disease involving the skin, the joints and the vascular compartment. The mechanisms linking inflammation in the skin and joints and in the vascular walls are poorly understood. One hypothesis for the increase in vascular inflammation observed in patients with psoriasis involves circulating pro-inflammatory cytokines. Patients with psoriasis have an increase in serum levels of tumor necrosis factor alpha (TNF-alpha), Interleukin-17 (IL-17), IL-22, IL-6 as well as a the chemokine S100A913. It is possible that one of those cytokines/chemokine induces vascular inflammation in the vascular compartment. The purpose of this cross sectional retrospective study is to highlight the correlation between vascular wall inflammation using 18F-2-fluoro-2-deoxy-D-glucose - Positron Emission Tomography (FDG-PET) fluorodeoxyglucose technology and pro-inflammatory cytokines/chemokine.

DETAILED DESCRIPTION:
Baseline frozen serum samples will be identified from the 107 enrolled Inno-6025 (Abbvie A13-935) (ClinicalTrials.gov Identifier NCT01722214) patients who also underwent a pre-adalimumab FDG-PET scan for the study. Serum cytokine and chemokine levels in these samples will be measured; IL-17 and IL-22 using the Singulex immunoassay platform, and S100A9, IL-6 and TNF alpha using multiplex ELISA. Vascular inflammation will be measured as the target to background ratio (TBR) in the ascending aorta using PET-scan technology. Correlation analyses will be performed between serum levels of cytokines and a chemokine and vascular inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has plaque psoriasis.
2. Patient has at least a 6 month history of plaque psoriasis.
3. Patient has a Body Surface Area (BSA) covered with psoriasis of 5% or more at Day 0.
4. Patient is a candidate for systemic therapy.
5. Patient is male or female, 18 to 80 years of age at time of consent.
6. Patient's weight at screening is a maximum of 180 kg.
7. Patient using medication to control angina, hypertension, serum lipids and any medication that can have an effect on inflammation must be on a stable dose for at least 8 weeks before Day 0.
8. Patient has an ascending aorta atherosclerotic plaque inflammation target-to-background ratio of 1.6 or more as determined by 18-FDG uptake measured by PET scanning.
9. Patient or patient's partner has been in a menopausal state for at least a year, is surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation or vasectomy), is clinically diagnosed infertile, has a same-sex partner, is abstinent, or is willing to use effective contraceptive method for at least 30 days before Day 0 and at least 6 months after the last study drug administration. Effective contraceptive methods are:

   1. Barrier methods such as condom, sponge or diaphragm combined with spermicide in foam, gel or cream;
   2. Hormonal contraception (oral, intramuscular, implant or transdermal) which include Depo-Provera, Evra and Nuvaring;
   3. Intrauterine device (IUD);
10. Female patients of childbearing potential must have a negative serum pregnancy test at the Screening visit.
11. Patient is judged to be in good general health as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination, and Chest X-Ray (CXR) performed at Screening.
12. Patient will be evaluated for latent TB infection with a purified protein derivative (PPD) or a Quantiferon Gold test and CXR. Patient who demonstrates evidence of latent TB infection (either PPD more than or equal to 5 mm of induration or positive Quantiferon Gold, irrespective of Bacillus Calmette-Guerin (BCG) vaccination status and negative CXR findings for active TB, and/or suspicious CXR findings) will not be allowed to participate in the study.
13. Patient must be able and willing to provide written informed consent and comply with the requirements of this study protocol.
14. Patient must be able and willing to self-administer subcutaneous (SC) injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

1. Patient has spontaneously improving or rapidly deteriorating plaque psoriasis.
2. Patient has other active infections (bacterial, fungal or viral) or skin diseases or skin infections (bacterial, fungal, or viral) that may interfere with evaluation of psoriasis or with patient's safety.
3. Patient has a history of an allergic reaction or significant sensitivity to constituents of study drug, including latex (a component of the pre-filled syringe).
4. Patient has used a non-biological systemic therapy for the treatment of psoriasis less than 30 days before Day 0.
5. Patient has used an investigational chemical or biological agent less than 30 days or 5 half-lives prior to the Day 0 visit (whichever is longer).
6. Patient has used a biological therapy for the treatment of psoriasis less than 90 days before day 0.
7. Patient has used a systemic immunosuppressor (eg. Azathioprine, 6-mercaptopurine) less than 30 days before Day 0.
8. Patient is taking or requires oral or injectable corticosteroids during the study. Inhaled corticosteroids for stable medical conditions are allowed.
9. Patient has used a topical treatment for psoriasis or has used phototherapy within the last 2 weeks prior to Day 0 (at the exception of low potency topical corticosteroids for groin, genitals, face, inframammary area, palms and soles).
10. Patient has received Anakinra/Kineret within the last 2 weeks prior to the Day 0 visit or is likely to receive Anakinra/Kineret during the course of the study
11. Patient has a poorly controlled medical condition, such as uncontrolled diabetes, documented history of recurrent infections, unstable ischemic heart disease, class III or IV (New York Heart Association Functional Classification; NYHA) congestive heart failure, an ejection fraction of less than 30%, recent stroke (within the past 3 months), chronic leg ulcer or any other condition which, in the opinion of the investigator, would put the patient at risk if participating in the study.
12. Patient has had a myocardial infarction or has been hospitalized for a cardiac condition within the past 12 weeks.
13. Patient has a history of acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft, carotid endarterectomy, stent installation or carotid revascularization within 12 weeks of Day 0.
14. Patient has had a percutaneous coronary intervention in the past 12 months.
15. Patient plans for a change in medical treatment for angina, serum lipids, hypertension or any other medication that can have a significant effect on inflammation during the course of the study.
16. Patient has history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease (e.g. optic neuritis, visual disturbance, gait disorder/ataxia, facial paresis, apraxia).
17. Patient has history of cancer or lymphoproliferative disease other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
18. Patient has a history of listeriosis, treated or untreated Tuberculosis (TB), persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives within 30 days prior to the Day 0 visit or oral anti-infectives within 14 days prior to the Day 0 visit.
19. Patient has received a live attenuated vaccine 28 days or less before Day 0 or plan to receive a live attenuated vaccine during the study and up to 4 months after the last study drug administration..
20. Patient with hepatitis B or hepatitis C viral infection
21. Patient with any of the following: hemoglobin ≤ 10 g/L, white blood cell count ≤ 3.0 X 109/L, platelet count ≤130 X 10^9/L, alanine transaminase (ALT) ≥ 2 times the upper limit of normal, aspartate transaminase (AST) ≥ 3 times the upper normal limit, total bilirubin ≥ 2 times the upper normal limit or creatinine ≥ 150 µmol/L.
22. Patient currently uses or plans to use anti-retroviral therapy at any time during the study.
23. Patient is known to have immune deficiency or is immunocompromised.
24. Female patient who is pregnant or breast-feeding or considering becoming pregnant during the study or for 6 months after the last dose of study medication.
25. Patient has a history of clinically significant drug or alcohol abuse in the last year.
26. Patient who plans to travel in an area where tuberculosis is endemic during the study and up to 4 months after the last study drug administration.
27. Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously enrolled in the Inno-6025 Trial (ClinicalTrials.gov Identifier NCT01722214)
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Correlation between serum cytokine levels (pg/mL) and TBR in the ascending aorta. | Baseline
  Correlation between serum levels of various cytokines including TNF alpha, IL-17, IL-22 and IL-6 and vascular inflammation measured as TBR using FDG-PET in patients with moderate to severe psoriasis

SECONDARY OUTCOMES:
Correlation between a serum chemokine (S100A9 (pg/mL)) levels and TBR in the ascending aorta. | Baseline
  Correlation between serum levels of a chemokine (S100A9) and vascular inflammation measured as TBR using FDG-PET in patients with moderate to severe psoriasis

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research
Locations (4):
- Canada (4):
  - Lynderm Research, Markham, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Clinique Dre Isabelle Delorme, Drummondville, Quebec
  - Innovaderm Research, Montreal, Quebec